CLINICAL TRIAL: NCT02092350
Title: A Phase II/III Randomized Clinical Trial to Study the Efficacy and Safety of the Combination Regimen of MK-5172 and MK-8742 in Subjects With Chronic Hepatitis C Virus Infection and Chronic Kidney Disease
Brief Title: Safety and Efficacy of Grazoprevir (MK-5172) + Elbasvir (MK-8742) in Participants With Chronic Hepatitis C and Chronic Kidney Disease (MK-5172-052)
Acronym: C-SURFER
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5172-052; 2013-003858-25 (EudraCT Number)
Record Dates: First submitted 2014-03-17; First posted 2014-03-20 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir; elbasvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Immediate Treatment (Experimental): Participants receive grazoprevir 100 mg tablet, orally, once per day (QD) + elbasvir 50 mg tablet, orally, QD, for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir
- Deferred Treatment (Experimental): Participants receive placebos to both grazoprevir and elbasvir for 12 weeks, and after a 4-week break, grazoprevir 100 mg tablet, orally, QD + elbasvir 50 mg tablet, orally, QD for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Placebo to Grazoprevir; Drug: Placebo to Elbasvir
- Intensive PK (Experimental): Participants receive grazoprevir 100 mg tablet, orally, QD + elbasvir 50 mg tablet, orally, QD for 12 weeks with intensive PK testing.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir

INTERVENTIONS:
Drug: Grazoprevir — Grazoprevir 100 mg tablet
  Other Names: MK-5172
Drug: Elbasvir — Elbasvir 50 mg tablet
  Other Names: MK-8742
Drug: Placebo to Grazoprevir — Placebo tablet matched to grazoprevir
  Arms: Deferred Treatment
Drug: Placebo to Elbasvir — Placebo tablet matched to elbasvir
  Arms: Deferred Treatment

SUMMARY:
This study will evaluate the safety and efficacy of combination treatment with grazoprevir (MK-5172) + elbasvir (MK-8742) for cirrhotic and non-cirrhotic participants with chronic Genotype 1 (GT1) hepatitis C virus (HCV) infection and chronic kidney disease (CKD). The primary study hypothesis is that the proportion of HCV GT1-infected CKD participants within the Immediate Treatment and Intensive Pharmacokinetics (PK) groups achieving a sustained viral response 12 weeks after the end of all study treatment (SVR12) will be >45%.

ELIGIBILITY:
Inclusion Criteria:

* Documented chronic (at least 6 months) HCV GT 1 infection (with no evidence of mixed genotypes or genotype that cannot be assigned a type)
* Evidence or no evidence of liver cirrhosis based on one of the following:
* Liver biopsy performed within 24 months of Day 1 (if participant is cirrhotic then there is no time restriction on biopsy)
* Fibroscan performed within 12 months of Day 1 of this study
* Fibrosure™ (Fibrotest™) plus aspartate aminotransferase to platelet Ratio Index [APRI] obtained during the screening period)
* Has HCV status that is one of the following:
* Treatment naïve
* Prior interferon or pegylated interferon with or without ribavarin failures (null responder, partial responder, or relapser)
* Intolerant to prior interferon or pegylated intereferon with or without ribavarin regimen
* Chronic kidney disease (defined as glomerular filtration rate [eGFR] <=29) non-dialysis dependent or on hemodialysis for at least 3 months, including individuals awaiting kidney transplant and those with failed kidney transplants but no longer on immunosuppressant therapy)
* Female participant of reproductive potential must agree to remain abstinent or use (or have their partner use) 2 acceptable methods of contraception from at least 2 weeks prior to Day 1 through 14 days after the last dose of study drugs, or longer if dictated by local regulations

Exclusion Criteria:

* Evidence of decompensated liver disease
* On peritoneal dialysis for management of kidney disease
* Co-infection with hepatitis B virus or human immunodeficiency virus (HIV)
* History of malignancy <=5 years prior to signing informed consent
* Clinical diagnosis of substance abuse
* Pregnant, breast-feeding, expecting to conceive or donate eggs, or donate sperm from Day 1 through 14 days after the last study dose, or longer if dictated by local regulations
* Organ transplant (including hematopoietic stem cell transplant) other than kidney, cornea, and hair
* Conditions requiring, or likely to require, chronic systemic administration of corticosteroids during the course of the trial
* Uncontrolled or poorly controlled hypertension
* Significant cardiovascular disorder (e.g. myocardial infarction or unstable angina) or cardiovascular procedure within 3 months prior to signing informed consent
* New or worsening signs or symptoms of congestive heart failure within 3 months of signing informed consent
* Severe active peripheral vascular disease
* Recent (within 3 months prior to signing informed consent) episode or recurrence of stroke, transient ischemic attack (TIA) or neurological disorder, including but not limited to seizures
* Evidence or history of chronic hepatitis not caused by HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2014-03-17 (Actual); Primary Completion 2015-03-11 (Actual); Study Completion 2015-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Roth D, Nelson DR, Bruchfeld A, Liapakis A, Silva M, Monsour H Jr, Martin P, Pol S, Londono MC, Hassanein T, Zamor PJ, Zuckerman E, Wan S, Jackson B, Nguyen BY, Robertson M, Barr E, Wahl J, Greaves W. Grazoprevir plus elbasvir in treatment-naive and treatment-experienced patients with hepatitis C virus genotype 1 infection and stage 4-5 chronic kidney disease (the C-SURFER study): a combination phase 3 study. Lancet. 2015 Oct 17;386(10003):1537-45. doi: 10.1016/S0140-6736(15)00349-9. Epub 2015 Oct 5. PMID 26456905
- [Result] Bruchfeld A, Roth D, Martin P, Nelson DR, Pol S, Londono MC, Monsour H Jr, Silva M, Hwang P, Arduino JM, Robertson M, Nguyen BY, Wahl J, Barr E, Greaves W. Elbasvir plus grazoprevir in patients with hepatitis C virus infection and stage 4-5 chronic kidney disease: clinical, virological, and health-related quality-of-life outcomes from a phase 3, multicentre, randomised, double-blind, placebo-controlled trial. Lancet Gastroenterol Hepatol. 2017 Aug;2(8):585-594. doi: 10.1016/S2468-1253(17)30116-4. Epub 2017 May 30. PMID 28576451
- [Derived] Prabhu AR, Rao IR, Nagaraju SP, Rajwar E, Venkatesh BT, Nair N S, Pai G, Reddy NP, Suvarna D. Interventions for dialysis patients with hepatitis C virus (HCV) infection. Cochrane Database Syst Rev. 2023 Apr 25;4(4):CD007003. doi: 10.1002/14651858.CD007003.pub3. PMID 37096802
- [Derived] Caro L, Wenning L, Feng HP, Guo Z, Du L, Bhagunde P, Fandozzi C, Panebianco D, Marshall WL, Butterton JR, Iwamoto M, Yeh WW. Pharmacokinetics of elbasvir and grazoprevir in subjects with end-stage renal disease or severe renal impairment. Eur J Clin Pharmacol. 2019 May;75(5):665-675. doi: 10.1007/s00228-018-2585-3. Epub 2019 Jan 25. PMID 30680407
- [Derived] Reau N, Robertson MN, Feng HP, Caro L, Yeh WW, Nguyen BT, Wahl J, Barr E, Hwang P, Klopfer SO. Concomitant proton pump inhibitor use does not reduce the efficacy of elbasvir/grazoprevir: A pooled analysis of 1,322 patients with hepatitis C infection. Hepatol Commun. 2017 Aug 22;1(8):757-764. doi: 10.1002/hep4.1081. eCollection 2017 Oct. PMID 29404492
- [Derived] Jacobson IM, Lawitz E, Kwo PY, Hezode C, Peng CY, Howe AYM, Hwang P, Wahl J, Robertson M, Barr E, Haber BA. Safety and Efficacy of Elbasvir/Grazoprevir in Patients With Hepatitis C Virus Infection and Compensated Cirrhosis: An Integrated Analysis. Gastroenterology. 2017 May;152(6):1372-1382.e2. doi: 10.1053/j.gastro.2017.01.050. Epub 2017 Feb 11. PMID 28193518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multi-site study enrolled adult, male and female participants with hepatitis C virus (HCV) genotype (GT) 1 with chronic kidney disease (CKD).
Pre-assignment Details: The screening period lasted for up to 60 days.
Groups:
- Immediate Treatment + Intensive PK: Participants received grazoprevir (GZR) 100 mg tablet + elbasvir (EBR) 50 mg tablet once daily (q.d.) by mouth for 12 weeks, followed by a 24-week follow-up period. A subset of participants also underwent intensive pharmacokinetics (PK) testing.
- Deferred Treatment: Participants received placebo to GZR and EBR q.d. by mouth for 12 weeks. Then, after a 4-week drug-free period, participants received a fixed dose combination (FDC) tablet containing GZR 100 mg + EBR 50 mg tablet q.d. by mouth for 12 weeks, followed by a 24-week follow-up period.
Period: Overall Study
Arm/Group | Immediate Treatment + Intensive PK | Deferred Treatment
Started | 123 | 114
Completed | 113 | 102
Not Completed | 10 | 12
Not completed — Adverse Event | 0 | 3
Not completed — Death | 2 | 5
Not completed — Lost to Follow-up | 3 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Screen Failure | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Immediate Treatment + Intensive PK: Participants received GZR 100 mg tablet + EBR 50 mg tablet q.d. by mouth for 12 weeks, followed by a 24-week follow-up period. A subset of participants also underwent intensive PK testing.
- Deferred Treatment: Participants received placebo to GZR and EBR q.d. by mouth for 12 weeks. Then, after a 4-week drug-free period, participants received a FDC tablet containing GZR 100 mg + EBR 50 mg tablet q.d. by mouth for 12 weeks, followed by a 24-week follow-up period.
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment + Intensive PK | Deferred Treatment | Total
Number analyzed (Participants) | 123 | 114 | 237
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (9.0) | 55.2 (10.0) | 55.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 33 | 63
  Male | 93 | 81 | 174

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Completing Study Therapy (SVR12)
Description: SVR12 was defined as hepatitis C virus (HCV) ribonucleic acid (RNA) lower than the limit of quantification (LLoQ) 12 weeks after completing study therapy. HCV RNA was measured using the COBAS™ AmpliPrep/COBAS™ Taqman™ HCV Test, v2.0®, which has a LLoQ of 15 IU/mL.
Time Frame: Week 24 (Immediate Treatment + Intensive PK) or Week 40 (Deferred Treatment)
Population: The modified Full Analysis set (mFAS) includes all participants receiving ≥1 dose of drug and without missing data due to death or early discontinuation from study therapy for reasons unrelated to response to HCV treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Immediate Treatment + Intensive PK | Deferred Treatment
Number analyzed (Participants) | 116 | 99
Percentage of participants | 99.1 [95.3 to 100.0] | 98.0 [92.9 to 99.8]
Statistical Analysis 1: Comparison: Immediate Treatment + Intensive PK; The primary hypothesis was that the SVR12 rate in the Immediate Treatment plus Intensive PK arm would be >45%; Test type: Superiority or Other; p = 0.001, One-sided exact test

2. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE) During the Initial Treatment and 14-day Follow-up Periods
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. This analysis includes the Immediate Treatment + Intensive PK group and the placebo treatment period for the Deferred Treatment group.
Time Frame: Up to Week 14
Population: The All Participants as Treated (APaT) population includes all enrolled participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Immediate Treatment + Intensive PK | Deferred Treatment
Number analyzed (Participants) | 122 | 113
Participants | 93 | 96

3. Primary Outcome: Number of Participants Discontinuing Study Drug Due to AEs During the Initial Treatment Period
Description: as for outcome 2
Time Frame: Up to Week 12
Population: The APaT population includes all enrolled participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Immediate Treatment + Intensive PK | Deferred Treatment
Number analyzed (Participants) | 122 | 113
Participants | 0 | 5

4. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks After Completing Study Therapy (SVR24)
Description: SVR24 was defined as HCV RNA <LLoQ 24 weeks after completing study therapy. HCV RNA was measured using the COBAS™ AmpliPrep/COBAS™ Taqman™ HCV Test, v2.0®, which has a LLoQ of 15 IU/mL.
Time Frame: Week 36 (Immediate Treatment + Intensive PK) or Week 52 (Deferred Treatment)
Population: The mFAS includes all participants receiving ≥1 dose of drug and without missing data due to death or early discontinuation from study therapy for reasons unrelated to response to HCV treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Deferred Treatment Group: Participants received placebo to GZR and EBR q.d. by mouth for 12 weeks. Then, after a 4-week drug-free period, participants received a FDC tablet containing GZR 100 mg + EBR 50 mg tablet q.d. by mouth for 12 weeks, followed by a 24-week follow-up period.
Arm/Group | Immediate Treatment + Intensive PK | Deferred Treatment Group
Number analyzed (Participants) | 114 | 99
Percentage of participants | 97.4 [92.5 to 99.5] | 98.0 [92.9 to 99.8]

5. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 Weeks After Completing Study Therapy (SVR4)
Description: SVR4 was defined as HCV RNA <LLoQ 4 weeks after completing study therapy. HCV RNA was measured using the COBAS™ AmpliPrep/COBAS™ Taqman™ HCV Test, v2.0®, which has a LLoQ of 15 IU/mL.
Time Frame: Week 16 (Immediate Treatment + Intensive PK) or Week 32 (Deferred Treatment)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Immediate Treatment + Intensive PK | Deferred Treatment Group
Number analyzed (Participants) | 118 | 101
Percentage of participants | 100.00 [96.9 to 100.0] | 99.0 [94.6 to 100.0]

ADVERSE EVENTS:
Time Frame: Immediate Treatment + Intensive PK: up to Week 36; Deferred Treatment GZR Placebo + EBR Placebo: up to Week 16; Deferred Treatment GZR 100 mg + EBR 50 mg: Week 16 to up to Week 52.
Description: AE data is presented for APaT (all participants receiving ≥1 dose of study drug).
Groups:
- Deferred Treatment: GZR Placebo + EBR Placebo 12 Weeks: Participants received placebo to GZR and EBR q.d. by mouth for 12 weeks, followed by a 4-week drug-free period.
- Deferred Treatment: GZR 100 mg + EBR 50 mg 12 Weeks: Participants received a FDC tablet containing GZR 100 mg + EBR 50 mg q.d. by mouth for 12 weeks, followed by a 24-week follow-up period.
Arm/Group | Immediate Treatment + Intensive PK | Deferred Treatment: GZR Placebo + EBR Placebo 12 Weeks | Deferred Treatment: GZR 100 mg + EBR 50 mg 12 Weeks
Serious Adverse Events (participants affected / at risk) | 30/122 | 22/113 | 25/102
Other Adverse Events (participants affected / at risk) | 67/122 | 68/113 | 39/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Treatment + Intensive PK (N=122) | Deferred Treatment: GZR Placebo + EBR Placebo 12 Weeks (N=113) | Deferred Treatment: GZR 100 mg + EBR 50 mg 12 Weeks (N=102)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 2 (3)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Citrobacter sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterobacter sepsis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected fistula (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Dialysis related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Genital injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Cryoglobulinaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nocardiosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mediastinal effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Treatment + Intensive PK (N=122) | Deferred Treatment: GZR Placebo + EBR Placebo 12 Weeks (N=113) | Deferred Treatment: GZR 100 mg + EBR 50 mg 12 Weeks (N=102)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 6 (6) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 10 (13) | 3 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 8 (8) | 6 (7) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 15 (22) | 5 (6)
Nausea (Gastrointestinal disorders) | 18 (24) | 18 (21) | 11 (12)
Vomiting (Gastrointestinal disorders) | 9 (13) | 9 (11) | 7 (10)
Asthenia (General disorders) | 7 (9) | 6 (6) | 4 (4)
Fatigue (General disorders) | 13 (15) | 17 (17) | 10 (10)
Pyrexia (General disorders) | 6 (7) | 6 (6) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 7 (8) | 3 (3) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (9) | 2 (2)
Dizziness (Nervous system disorders) | 8 (9) | 18 (22) | 4 (4)
Headache (Nervous system disorders) | 23 (26) | 18 (23) | 7 (8)
Insomnia (Psychiatric disorders) | 10 (10) | 12 (12) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 2 (2) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 12 (12) | 1 (1)
Hypertension (Vascular disorders) | 7 (7) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.